CLINICAL TRIAL: NCT05305898
Title: MetCool ACS"- Metformin "Cooling" Effect on Metformin-naive Patients Treated With PCI Because of Acute Coronary Syndrome
Brief Title: "MetCool ACS"- Metformin "Cooling" Effect on Metformin-naive Patients Treated With PCI Because of Acute Coronary Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: ABM Industries (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MC-ACS01-2020; 2020-004962-21 (EudraCT Number)
Record Dates: First submitted 2022-02-17; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): Patients from "metformin group" will receive metformin 3 x 850 mg (after titration period) for 2 years (3 x 500 mg for first 6 weeks) with 6 months follow-up after treatment cessation.
  Interventions: Drug: Metformin
- No metformin group (No Intervention): Patients form "no metformin" group will be observed for 2 years and 6 months, which cover the same period like for patients from metformin group.

INTERVENTIONS:
Drug: Metformin — Patients from "metformin group" will receive metformin 3 x 850 mg (after titration period) for 2 years (3 x 500 mg for first 6 weeks) with 6 months follow-up after treatment cessation.
  Arms: Metformin group

SUMMARY:
The aim of the study is the evaluation of the effect of metformin among the patients without diabetes, on the incidence of reintervention, unplanned revascularization, after full percutaneous coronary revascularization as a result of the first episode of the acute coronary syndrome (ACS).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* ACS, according to the current definition of the European Society of Cardiology, treated with percutaneous coronary intervention with drug eluting stent implantation
* Occupation and place of residence not causing difficulties in participating in control visits
* Uncomplicated course of the disease (ACS) as assessed by the treating physician
* Negative history of diabetes
* Not taking any hypoglycaemic drugs prior to hospitalization immediately or within the last 6 months
* HbA1c< 6,5% (assessment during hospitalization)
* Written consent to participate in the study

Exclusion Criteria:

* Significant valve disease confirmed by ECHO
* Previous CABG
* NYHA IV during hospitalization
* Chronic kidney disease with GFR <60 ml / min / 1.73 m2 according to MDRD
* ALT three times above normal according to laboratory criteria
* Serious co-morbidities and estimated survival less than 2.5 years, as assessed by the treating physician
* Known gastrointestinal disease that may potentially be responsible for the intolerance to metformin (e.g. inflammatory bowel disease, gastro-oesophageal reflux disease)
* Known potential difficulties in cooperation with patients (dementia, mental disorders, distance from the place of residence, if considered potentially problematic, alcoholism)
* Hypersensitivity to metformin
* Pregnancy and breastfeeding
* Patient participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Need for unscheduled PCI or CABG after successful final stage of revascularization due to ACS within a 30-month follow-up period | through study completion, an average of 5 years
  Number of patients who needs an unscheduled PCI or CABG after successful final stage of revascularization due to ACS within a 30-month follow-up period

SECONDARY OUTCOMES:
Death from cardiac causes after successful final stage of revascularization due to ACS within 30 months of follow-up | through study completion, an average of 5 years
  Number of deaths from cardiac causes after successful final stage of revascularization due to ACS within 30 months of follow-up
All-cause death following successful final stage revascularization for ACS within a 30-month follow-up period | through study completion, an average of 5 years
  Number of all-cause deaths following successful final stage revascularization for ACS within a 30-month follow-up period
Non-fatal myocardial infarction after successful final stage of revascularization due to ACS within 30 months of follow-up | through study completion, an average of 5 years
  Number of non-fatal myocardial infarctions after successful final stage of revascularization due to ACS within 30 months of follow-up
Non-fatal stroke after successful final stage of revascularization due to ACS within 30 months of follow-up | through study completion, an average of 5 years
  Number of non-fatal strokes after successful final stage of revascularization due to ACS within 30

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Gierelak, Principal Investigator — Military Institute of Medicine
Locations (14):
- Poland (14):
  - Oddział Kardiologii Szpitala św. Rafała, Krakow, Lesser Poland Voivodeship
  - Wielospecjalistyczny Szpital Wojewódzki w Gorzowie Wielkopolskim, Gorzów Wielkopolski, Lubusz Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - Kluczborskie Centrum Kardiologii, Kluczbork, Opole Voivodeship
  - Centrum Kardiologii Scanmed w Bielsku Podlaskim, Bielsk Podlaski, Podlaskie Voivodeship
  - Chorzowskie Centrum Kardiologii, Chorzów, Silesian Voivodeship
  - Raciborskie Centrum Medyczne, Racibórz, Silesian Voivodeship
  - Sosnowieckie Centrum Kardiologii, Sosnowiec, Silesian Voivodeship
  - Centrum Kardiologii Scanmed w Ełku, Ełk, Warmian-Masurian Voivodeship
  - Centrum Kardiologii Scanmed w Iławie, Iława, Warmian-Masurian Voivodeship
  - Centrum Kardiologii Scanmed w Szczecinku, Szczecinek, West Pomeranian Voivodeship
  - Centrum Kardiologii Scanmed w Kutnie, Kutno, Łódź Voivodeship
  - Centrum Kardiologii Scanmed w Tomaszowie Mazowieckim, Tomaszów Mazowiecki, Łódź Voivodeship
  - Częstochowskie Centrum Kardiologii, Częstochowa, Śląske

IPD SHARING:
Plan to Share IPD: Undecided